CLINICAL TRIAL: NCT02207153
Title: Risk Assessment by Cardiovascular Biomarkers in Chronic Dialysis Patients
Acronym: RACE
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: EKNZ 2014-210
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Endstage Renal Disease
Keywords: Chronic Hemodialysis; Chronic Peritoneal Dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — At the beginning and the end of the dialysis session, at the time of the monthly routine blood tests additional venous blood samples will be collected. All draws will be performed after a three day interdialytic interval. Until the time of en bloc analysis the aliquots will be stored at -80°. All study data and blood samples will be stored for 10 years after study termination, for the future assessment of novel cardiovascular biomarkers. The stored blood samples will be anonymised and only labelled by a barcode. This barcode be unambiguously linked to the study ID code for the individual patient. There will be no direct link between the original participant details and the blood sample bar code.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic Hemodialysis: Initiation of chronic hemodialysis or currently undergoing chronic hemodialysis at one of the study centres
- Peritoneal Dialysis: Initiation of chronic peritoneal dialysis or currently undergoing chronic peritoneal dialysis at one of the study centres

SUMMARY:
Patients undergoing chronic dialysis are at a substantially increased risk of cardiac death. The reasons for this excess cardiovascular mortality are only partly understood. Classical complicated artherosclerotic disease does not appear to be the primary cause of cardiac death in chronic dialysis patients. In fact, the predictive potential of classic cardiovascular risk factors such as hypertension, obesity and hyperlipidemia appears to be reduced in dialysis. In contrast, in a series of pilot studies we found cardiac biomarkers to adequately reflect dialysis induced myocardial stunning, progressive cardiovascular disease, and the risk of death.

To extend and corroborate these results, we are planning a large, prospective, observational study enrolling unselected hemo- and peritoneal dialysis patients. The proposed study, its power calculation and hypotheses are based on our pilot studies

DETAILED DESCRIPTION:
Eligible patients will be identified through the clinical care team by undergoing chronic dialysis at one of the study centres. Dialysis patients will be initially approached during a routine dialysis session by a member of the clinical team to discuss the study and a participant information sheet will be provided. A minimum of 2 days after the provision of the participant information sheet, the clinical team will inform the research team about the patients who are interested in this study. Potential participants will be re-approached in person by a trained research physician to determine whether they are willing to participate in the study. If they are interested, the information sheet will be discussed with them and any questions will be answered. The investigators will explain the nature of the study, its purpose, the procedures involved, the expected duration, the potential risks and benefits and any discomfort it may entail to each potential participant. Each participant will be informed that the participation in the study is voluntary and that he/she may withdraw from the study at any time and that withdrawal of consent will not affect his/her subsequent medical assistance and treatment.

All potential study participants will be provided with a participant information sheet and a consent form describing the study and providing sufficient information for the participant to make an informed decision about their participation in the study.

The participant will be given a copy of the signed document. The consent form must also be signed and dated by the investigator (or his designee) and it will be retained as part of the study records. After consent is obtained, the participant will be allocated an unique study identification (ID) code.

Patients are free to discontinue their participation in the study at any time, without having to give a reason for their withdrawal.

Patient exposure will be censored for discontinuation of dialysis because of regaining renal function or patient's wish, study withdrawal and transfer of the patient to a non-participating dialysis unit. Patients undergoing renal transplantation during the observational period will not be censored, but will be reassessed 3 and 6 months after transplantation.

First, written informed consent will be obtained from the patient. After we have obtained informed consent patients will undergo their standard three times weekly hemodialysis sessions or their daily peritoneal dialysis session. At the time of enrolment into the trial all patients will undergo a detailed clinical assessment including a medical history and a physical examination. At the beginning and the end of the dialysis session, at the time of the monthly routine blood tests additional venous blood samples will be collected. Serial assessments will be performed in 6 monthly intervals until the enrollment target has been met. After reaching the enrollment target the observational period will continue for another year.

ELIGIBILITY:
Inclusion Criteria:

- Age ≥18 years

* Initiation of chronic hemodialysis or currently undergoing chronic hemodialysis at one of the study centres
* Initiation of chronic peritoneal dialysis or currently undergoing chronic peritoneal dialysis at one of the study centres
* Written informed consent

Exclusion Criteria:

* Age < 18 years
* No written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data of patients undergoing chronic hemodialysis and peritoneal dialysis will be analysed overall (RACE-Dial) and separately in the two substudies, RACE-HD and RACE-PD.
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Cardiac death | Weekly
  Cardiac death will be defined as death due to:
  * coronary artery disease
  * heart failure
  * arrhythmias
  * sudden death
  * or other heart diseases
  Sudden deaths will operationally be defined as witnessed and unwitnessed unexpected deaths, with a preceding duration of symptoms less than 24 hours for witnessed deaths, and less than the interval since the last dialysis session for unwitnessed deaths.

SECONDARY OUTCOMES:
All Cause Mortality | Weekly
  All Cause Mortality

OTHER OUTCOMES:
Combined cardiac endpoint | weekly
  acute myocardial infarction, acute heart failure hospitalisations and cardiac death

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Breidthardt, PD Dr, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Background] Breidthardt T, Kalbermatter S, Socrates T, Noveanu M, Klima T, Mebazaa A, Mueller C, Kiss D. Increasing B-type natriuretic peptide levels predict mortality in unselected haemodialysis patients. Eur J Heart Fail. 2011 Aug;13(8):860-7. doi: 10.1093/eurjhf/hfr057. Epub 2011 May 30. PMID 21628312
- [Background] Breidthardt T, Burton JO, Odudu A, Eldehni MT, Jefferies HJ, McIntyre CW. Troponin T for the detection of dialysis-induced myocardial stunning in hemodialysis patients. Clin J Am Soc Nephrol. 2012 Aug;7(8):1285-92. doi: 10.2215/CJN.00460112. Epub 2012 Jul 19. PMID 22822013
- [Background] Breidthardt T, Moser-Bucher CN, Praehauser C, Garzoni D, Bachler K, Steiger J, Dickenmann M, Mayr M. Morbidity and mortality on chronic haemodialysis: a 10-year Swiss single centre analysis. Swiss Med Wkly. 2011 Feb 3;141:w13150. doi: 10.4414/smw.2011.13150. eCollection 2011. PMID 21328099
- [Background] Breidthardt T, Burton JO, Odudu A, Eldehni MT, Jefferies H, McIntyre CW. N-terminal Pro-B-type natriuretic peptide and its correlation to haemodialysis-induced myocardial stunning. Nephron Clin Pract. 2013;123(1-2):118-22. doi: 10.1159/000351190. Epub 2013 Jul 18. PMID 23880872
- [Background] Breidthardt T, McIntyre CW. Dialysis-induced myocardial stunning: the other side of the cardiorenal syndrome. Rev Cardiovasc Med. 2011;12(1):13-20. doi: 10.3909/ricm0585. PMID 21546884